CLINICAL TRIAL: NCT03575182
Title: Gait Retraining in Patients With Joint Hypermobility Syndrome/Hypermobile Ehlers Danlos Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USF-JHS/hEDS-062118
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Joint Hypermobility; Ehlers-Danlos Syndrome; Hyperextension Knees
MeSH Terms: conditions — Joint Instability; Ehlers-Danlos Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait retraining program (Experimental)
  Interventions: Other: Gait retraining program
- Physical therapy standard care (No Intervention)

INTERVENTIONS:
Other: Gait retraining program — Supervised gait retraining with verbal and real-time visual feedback.
  Arms: Gait retraining program

SUMMARY:
This study evaluates the efficacy of gait retraining with biofeedback in the treatment of neuromusculoskeletal symptoms in patients with Joint Hypermobility Syndrome/Hypermobile Ehlers Danlos Syndrome. Half of participants will participate in a gait retraining program, while the other half will continue standard care.

ELIGIBILITY:
Inclusion Criteria:

* Ehlers-Danlos Syndrome Hypermobile type as defined in the 2017 international Ehlers-Danlos Syndrome classification

Exclusion Criteria:

* Other heritable and acquired connective tissue disorders, autoimmune rheumatologic conditions, pregnancy, history of lower limb surgery, cardiovascular limitations, visual limitations.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Knee Joint Range of Motion | 4-5 weeks